CLINICAL TRIAL: NCT02825667
Title: Randomized Clinical Study on the Effectiveness of the Myofascial Therapy in the Treatment of the Hemophilic Arthropathy of Ankle
Brief Title: Effectiveness of the Myofascial Therapy in the Hemophilic Arthropathy of Ankle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Real Fundación Victoria Eugenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AnHe-Fascial
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Haemophilia
Keywords: Haemophilia; Ankle; Arthropathy; Pain; Range of motion; Myofascial techniques
MeSH Terms: conditions — Hemophilia A; Joint Diseases; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Patients included in this group will receive treatment over a period of three weeks, receiving 3 physiotherapy sessions lasting approximately 30 minutes each.
  The treatment program includes 8 maneuvers that must be administered bilaterally: maneuver longitudinal sliding on the fascial surface plant, maneuver induction of the plantar fascia, maneuver longitudinal surface sliding on the anterolateral compartment of the leg, induction maneuver ankle anterior compartment, maneuver pressure and sliding on the posterior region of the leg, technical release of the popliteal fascia, maneuver induction sural triceps, and lower extremity telescopic technique.
  Interventions: Other: Physiotherapy sessions
- Control group (No Intervention): Patients included in this group will not receive any physiotherapy treatment. However, will be evaluated under the same conditions that patients in the experimental group (pretreatment evaluation, post-treatment and follow-up).

INTERVENTIONS:
Other: Physiotherapy sessions — Physiotherapy by techniques myofascial therapy, in patients with ankle hemophilic arthropathy
  Arms: Experimental group

SUMMARY:
Randomized clinical trial to assess the efficacy of a treatment protocol applied fascial therapy in patients with hemophilic arthropathy ankle, oriented to know and describe the observed differences on the dependent variables: range of motion, pain and physical condition.

At the same time, the study will determine whether there are adverse effects or bleeding complications as a result of applied physiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B
* Adults patients
* Patients with hemophilic arthropathy of ankle diagnosed
* Patients in prophylactic treatment regimen or on demand treatment with concentrates of FVIII/FIX.

Exclusion Criteria:

* Patients without ambulation
* Patients diagnosed with other congenital coagulopathy (eg, Von Willebrand disease)
* Patients who have developed antibodies to FVIII / FIX (inhibitors)
* Patients with neurological or cognitive impairments that prevent understanding of questionnaires and test physical
* Patients that have not signed the informed consent document.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline bleeding frequency after treatment and at 5 months | Screening visit, within the first seven days after treatment and after five months follow-up visit
  Evaluation of the frequency of muscle and joint bleeds through registration. The frequency of bleeding of the ankle joint is measured with a registry given to patients at the beginning of the study.
Change from baseline joint pain of ankle after treatment and at 5 months | Screening visit, within the first seven days after treatment and after five months follow-up visit
  Change from joint pain of ankle during treatment and follow-up period at 5 months. The perception of ankle pain will be measured using visual analog scale (scale 0-10).
Change from baseline joint function after treatment and at 5 months | Screening visit, within the first seven days after treatment and after five months follow-up visit
  Change from joint health during treatment and follow-up period at 5 months. Measurement instrument: Haemophilia Joint Health Score (scale 0-20).
Change from baseline range of motion after treatment and at 5 months | Screening visit, within the first seven days after treatment and after five months follow-up visit
  Change from range of movement of ankle and knee during treatment and follow-up period at 5 months. The range of motion of the ankle joint will be measured using a universal goniometer, using the protocol for measuring joint motion described by Felipe Querol.
  Measurement instrument: universal goniometer with the protocol to measurement for patients with hemophilia

SECONDARY OUTCOMES:
Age | Screening visit
  Age of patients
Weight | Screening visit
  Weight of patients included in the study
Height | Screening visit
  Height of patients

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Real Fundación Victoria Eugenia

IPD SHARING:
Plan to Share IPD: No